CLINICAL TRIAL: NCT05073198
Title: The Effect of the Brochure Given to University Students on Testicular Cancer and Its Early Diagnosis on Health Beliefs and Testicular Self-Examination
Brief Title: The Effect of the Brochure on Testicular Self-Exam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, BUSRA ALTINEL, Principal Investigator dr, Selcuk University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20202002
Record Dates: First submitted 2021-09-19; First posted 2021-10-11 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-09

CONDITIONS: Testicular Cancer
Keywords: testicular cancer; screening; university student
MeSH Terms: conditions — Testicular Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment (Experimental): Giving educational brochures about testicular cancer and Testicular Self-Examination to the students in the experimental group
  Interventions: Other: Education brochure
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: Education brochure — In the content of the brochure about testicular cancer and CCTM prepared in line with the literature; It includes information such as the definition of testicular cancer, testicular cancer risk factors and symptoms, the importance of early diagnosis in testicular cancer, how CCTM is performed, and what to do in case of differences after the examination. Expert opinion was obtained from three faculty members (a professor from the Department of Urology, a professor in Public Health Nursing and a physician faculty member) regarding the content validity of the educational brochure created before the research.
  Arms: Experiment

SUMMARY:
This study aims to examine the effect of the educational brochure given to university students on testicular cancer and its early diagnosis on their health beliefs and self-examination; In non-randomized groups, pretest-posttest was conducted in a quasi-experimental design with control group. The research was carried out with students studying in the psychological counseling and guidance department of a state university in Turkey. The study group consisted of 92 students, 48 of which were experimental and 44 were control. Only the experimental group was given an educational brochure about testicular cancer and testicular self-examination. Data; Personal information form, testicular cancer and health beliefs scale about testicular self-examination were collected with the form for self-examination. In the evaluation of the data; Mann Whitney U, Wilcoxon and chi-square analyzes were performed.

ELIGIBILITY:
Inclusion Criteria:

* To study in the Department of Psychological Counseling and Guidance
* Studying in 3rd and 4th grade

Exclusion Criteria:

* Any previous diagnosis of cancer
* Having received previous training in Testicular Self Examination

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — testicular cancer is a type of cancer seen in men
Enrollment: 92 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2021-06-16 (Actual)

PRIMARY OUTCOMES:
rate of testicular self-exam | after 4 weeks
  After the training brochure given to the students, they are expected to do testicular examination on their own.

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes